CLINICAL TRIAL: NCT01292642
Title: Cognitive Behavioral Therapy and the Nicotine Transdermal Patch for Cannabis Dependence and Nicotine Dependence
Acronym: CBT-MJ-NIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Kevin P. Hill, MD, MHS, Instructor in Psychiatry, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-000927
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Results first posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Cannabis Dependence; Nicotine Dependence
Keywords: cognitive behavioral therapy; nicotine dependence; cannabis dependence; smoking cessation; nicotine replacement therapy
MeSH Terms: conditions — Marijuana Abuse; Tobacco Use Disorder; Smoking Cessation | interventions — Cognitive Behavioral Therapy; Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Cognitive behavioral therapy (CBT) plus transdermal patch nicotine replacement therapy (NRT) to treat co-occurring nicotine and cannabis dependence during a 10-week study.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — individual CBT once weekly, 50 minutes, for 10 weeks
Drug: Nicotine Replacement Therapy — 1. 21 mg patch for 6 weeks, 14 mg patch for 2 weeks, then 7 mg patch for 2 weeks
  2. 14 m g patch for 8 weeks, then 7 mg patch for 2 weeks
  Other Names: Nicotine Transdermal Patch

SUMMARY:
The investigators are conducting a Stage 1 pilot feasibility study at McLean Hospital to develop and refine a Cognitive Behavioral Therapy (CBT) intervention. The investigators aim to develop a feasible 10-week integrated CBT intervention for the treatment of concurrent marijuana dependence and nicotine dependence. The investigators hypothesize that the CBT intervention, in conjunction with Nicotine Replacement Therapy (NRT) in the form of a transdermal nicotine patch, will reduce the use of marijuana and nicotine.

DETAILED DESCRIPTION:
The investigators will conduct a Stage 1 pilot feasibility study at McLean Hospital to develop and refine a Cognitive Behavioral Therapy (CBT) intervention. Twelve subjects (50% female, ages 18-65) who meet Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) criteria for both marijuana and nicotine dependence and seek treatment to stop using both marijuana and tobacco will receive individual CBT aimed at treating both disorders, as well as Nicotine Replacement Therapy (NRT) in the form of a transdermal nicotine patch. Subjects will start with a 21-mg nicotine patch for 6 weeks, followed by a taper to a 14-mg nicotine patch for 2 weeks and, finally, a 7-mg nicotine patch for 2 weeks. Others will start with a 14-mg patch for 8 weeks followed by a 7-mg patch for 2 weeks. All participants will receive 10 weeks of 1-hour weekly CBT with an experienced clinician. Follow-up visits, scheduled at 4, 6, 8, and 10 weeks, will evaluate of the durability of treatment effects on drug use and psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-65 years
* current DSM-IV cannabis dependence
* current DSM-IV nicotine dependence
* express a desire to quit cannabis and nicotine use within the next 30 days
* daily use of ≥ 10 tobacco cigarettes
* for women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy and additional pregnancy tests at weeks 4 and 8
* Expired breath carbon monoxide (CO) determination is greater than or equal to 7 ppm over ambient values

Exclusion Criteria:

* Current diagnosis of other drug or alcohol dependence (other than cannabis or nicotine)
* recent (within 3 months) significant cardiac disease
* current serious psychiatric illness or history of psychosis, schizophrenia, bipolar type I disorder or significant current suicidal or homicidal thoughts
* current use of bupropion
* current NRT or other smoking cessation treatment
* current CBT or other behavioral treatments for cessation of marijuana or tobacco smoking
* current smokeless tobacco use
* inability to read or write in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Hill, MD, MHS, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Marijuana Treatment Project Research Group. Brief treatments for cannabis dependence: findings from a randomized multisite trial. J Consult Clin Psychol. 2004 Jun;72(3):455-66. doi: 10.1037/0022-006X.72.3.455. PMID 15279529
- [Background] Hill, K.P., and Chang, G. Cognitive Behavioral Therapy and Nicotine Replacement for Smoking Cessation in Psychiatric Outpatients with Major Depression. Addictive Disorders and Their Treatment, 6: 67-72, 2007.
- [Background] Hall SM, Munoz RF, Reus VI. Cognitive-behavioral intervention increases abstinence rates for depressive-history smokers. J Consult Clin Psychol. 1994 Feb;62(1):141-6. doi: 10.1037//0022-006x.62.1.141. PMID 8034816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via online and newspaper advertisements.
Pre-assignment Details: Four participants were determined to be ineligible due to significant active Axis I psychopathology other than nicotine or cannabis dependence, one was ineligible due to an active medical issue that was referred for treatment, and one was ineligible due to a positive urine toxicology screen for an illicit substance other than cannabis.
Period: Overall Study
Arm/Group | Treatment
Started | 12
Completed | 7
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Treatment: CBT plus NRT
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Use
Description: cigarettes per day
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: cigarettes/day
Groups:
- PostTreatment - Cigarettes Per Day: CBT plus NRT
Arm/Group | Baseline - Cigarettes Per Day | PostTreatment - Cigarettes Per Day
Number analyzed (Participants) | 7 | 7
cigarettes/day | 12.6 (4.9) | 2.1 (4.2)

2. Primary Outcome: Cannabis Use
Description: cannabis inhalations per day
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: cannabis inhalations/day
Groups:
- Baseline - Cannabis Inhalations Per Day: CBT plus NRT
Arm/Group | Baseline - Cannabis Inhalations Per Day | Post Treatment - Cannabis Inhalations Per Day
Number analyzed (Participants) | 7 | 7
cannabis inhalations/day | 10.0 (5.3) | 8.0 (5.3)

3. Secondary Outcome: Client Satisfaction Questionnaire (CSQ-8) at 10 Weeks
Description: The Client Satisfaction Questionnaire (CSQ-8) is a self-report instrument used to assess satisfaction with health services and it was used to assess participant satisfaction with the treatment during this 10 week study. Scores range from 8 - 32 with higher values indicating higher satisfaction.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 7
Scores on a scale | 30.6 (1.9)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
slightly more than one-third of participants did not complete treatment. The small sample size and relatively high proportion of treatment non-completers may limit our interpretation of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No